CLINICAL TRIAL: NCT04659603
Title: Open-label, Multi-cohort, Phase 2 Trial, Evaluating the Efficacy and Safety of Tusamitamab Ravtansine (SAR408701) Monotherapy and in Combination in Patients With CEACAM5-positive Advanced Solid Tumors
Brief Title: Tusamitamab Ravtansine Monotherapy and in Combination in Patients With CEACAM5-positive Advanced Solid Tumors
Acronym: CARMEN-BT01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision, the decision is not related to any safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT16432; U1111-1244-1644 (Registry Identifier: ICTRP); 2020-003096-18 (EudraCT Number)
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Metastatic; Pancreatic Carcinoma Metastatic
MeSH Terms: interventions — tusamitamab ravtansine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A metastatic breast cancer (mBC) (Experimental): tusamitamab ravtansine every 2 weeks administered via intravenous infusion (IV)
  Interventions: Drug: tusamitamab ravtansine
- Cohort B metastatic pancreatic adenocarcinoma (mPAC) (Experimental): tusamitamab ravtansine every 2 weeks administered via intravenous infusion (IV)
  Interventions: Drug: tusamitamab ravtansine
- Cohort C Metastatic pancreatic adenocarcinoma (mPAC) (Experimental): tusamitamab ravtansine every 2 weeks combined with gemcitabine on Day 1, Day 8 and Day 15 every 4 weeks administered via intravenous infusion (IV)
  Interventions: Drug: tusamitamab ravtansine; Drug: Gemcitabine

INTERVENTIONS:
Drug: tusamitamab ravtansine — Pharmaceutical form:Concentrated solution for IV;
  Route of administration: IV infusion
  Other Names: SAR408701
Drug: Gemcitabine — Pharmaceutical form: Lyophilized powder for reconstitution or as a solution for infusion;
  Route of administration: IV infusion
  Arms: Cohort C Metastatic pancreatic adenocarcinoma (mPAC)

SUMMARY:
Primary Objective:

* For Cohort A, Cohort B, and Cohort C Part 2: To assess the antitumor activity of tusamitamab ravtansine in metastatic breast cancer (mBC) and tusamitamab ravtansine monotherapy and in combination with gemcitabine in metastatic pancreatic adenocarcinoma (mPAC)
* For Cohort C Part 1: Confirmation of the recommended tusamitamab ravtansine dose when administered in combination with gemcitabine

Secondary Objectives:

* To assess the safety and tolerability of tusamitamab ravtansine administered as monotherapy and in combination with gemcitabine
* To assess other efficacy parameters of tusamitamab ravtansine administered as monotherapy and in combination with gemcitabine
* To assess the immunogenicity of tusamitamab ravtansine
* To assess the pharmacokinetics (PK) of tusamitamab ravtansine and gemcitabine when given in combination

DETAILED DESCRIPTION:
The expected duration of study intervention for participants may vary, based on progression date and the cohort; median expected duration of study per participant is estimated at 8 months for Cohort A/C and 6 months for Cohort B (up to 1 month for screening, a median of 4 or 2 months for treatment in Cohort A/C and Cohort B respectively, a median of 1 month for EOT, and follow-up visit 90 days after the last IMP administration).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age
* Participants with at least one measurable lesion according to the RECIST v1.1 criteria that has not been irradiated (ie, newly arising lesions in previously irradiated areas are accepted).
* Participants with ECOG performance status 0 to 1.
* Evidence of metastatic disease.
* Expression of CEACAM 5 by centrally assessed IHC assay.
* Male and female participants willing to comply with contraceptive use consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Cohort A: mBC

* Histological or cytologic diagnosis of breast cancer.
* Have received at least 2 prior cytotoxic chemotherapy regimens for non-TNBC tumor type or at least 1 for TNBC tumor type but not more than 4 in the locally recurrent or metastatic setting.

Cohorts B and C: mPAC

- Have confirmed diagnosis of pancreatic ductal adenocarcinoma.

Cohort B: mPAC:

- Have documented radiographic progression or documented intolerance after at least 1 prior systemic chemotherapy line which included either gemcitabine (or relapsed within 6 months of completion of gemcitabine adjuvant therapy) or a 5-fluorouracil based regimen (including capecitabine) but no more than 2 prior chemotherapy lines for locally advanced/metastatic disease.

Cohort C: mPAC

- Have documented radiographic progression or documented intolerance after 1st line fluoropyrimidine-containing chemotherapy (or relapsed within 6 months of completion of chemotherapy as adjuvant therapy) for locally advanced/metastatic disease.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Medical condition requiring concomitant administration of a medication with a narrow therapeutic window, that is metabolized by cytochrome P450 (CYP450), and for which a dose reduction cannot be considered.
* Medical conditions requiring concomitant administration of strong CYP3A inhibitor, unless it can be discontinued at least 2 weeks before the first administration of study intervention.
* Life expectancy less than 3 months.
* Untreated brain metastases or history of leptomeningeal disease.
* Significant concomitant illness
* History within the last 3 years of an invasive malignancy other than the one treated in this study, with the exception of resected/ablated basal or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix, or other local tumors considered cured by local treatment.
* History of known acquired immunodeficiency syndrome (AIDS) related illnesses or known human immunodeficiency virus (HIV) disease requiring antiretroviral treatment, or active hepatitis A, B or C infection.
* Non-resolution of any prior treatment-related toxicity to <Grade 2 according to NCI CTCAE v5.0, with the exception of alopecia, vitiligo, or active thyroiditis controlled with hormone replacement therapy (HRT).
* Unresolved corneal disorder or any previous corneal disorder considered by an ophthalmologist to predict higher risk of drug-induced keratopathy.
* Use of contact lenses. Participants using contact lenses who are not willing to stop wearing them for the duration of the study intervention are excluded.
* Concurrent treatment with any other anti cancer therapy.
* Washout period before the first administration of study intervention of less than 3 weeks or less than 5 times the half-life, whichever is shorter, for prior antitumor therapy (chemotherapy, targeted agents, immunotherapy and radiotherapy, or any investigational treatment).
* Any prior therapy targeting CEACAM5.
* Prior maytansinoid DM4 treatment (ADC).
* Any major surgery within the preceding 2 weeks of the first study intervention administration.
* Previous enrollment in this study or current participation in any other clinical study involving an investigational study treatment or any other type of medical research.
* Poor renal function
* Poor hepatic function
* Poor bone marrow function

Cohort C: mPAC

- Any previous systemic therapy with taxane or gemcitabine (for Cohort C only).

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2025-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (29):
- United States (3):
  - AdventHealth Orlando Site Number : 8400001, Orlando, Florida
  - Massachusetts General Hospital Site Number : 8400002, Boston, Massachusetts
  - University of Wisconsin Site Number : 8400004, Madison, Wisconsin
- Argentina (3):
  - Investigational Site Number : 0320003, Capital Federal, Buenos Aires
  - Investigational Site Number : 0320001, Pergamino, Buenos Aires
  - Investigational Site Number : 0320002, Rosario, Santa Fe Province
- Chile (3):
  - Investigational Site Number : 1520002, Temuco, La Araucanía
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
- Investigational Site Number : 3480003, Budapest, Hungary
- Netherlands (3):
  - Investigational Site Number : 5280002, Amsterdam
  - Investigational Site Number : 5280001, Rotterdam
  - Investigational Site Number : 5280003, Utrecht
- Russia (3):
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430004, Pushkin, Saint- Petersburg
  - Investigational Site Number : 6430002, Saint Petersburg
- South Korea (3):
  - Investigational Site Number : 4100003, Goyang-si, Gyeonggi-do
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
- Spain (3):
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240002, Majadahonda, Madrid
  - Investigational Site Number : 7240003, Madrid, Madrid, Comunidad de
- Taiwan (3):
  - Investigational Site Number : 1580001, Taichung
  - Investigational Site Number : 1580002, Tainan
  - Investigational Site Number : 1580003, Taipei
- Turkey (Türkiye) (4):
  - Investigational Site Number : 7920003, Adana
  - Investigational Site Number : 7920004, Ankara
  - Investigational Site Number : 7920001, Istanbul
  - Investigational Site Number : 7920002, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT16432 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25192&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 31 centers in 10 countries. A total of 55 participants were screened from 29 March 2021 to 27 November 2023, of which 5 were screen failures. Screen failures were mainly due to not meeting the eligibility criteria.
Pre-assignment Details: Total 50 participants enrolled to receive tusamitamab ravtansine as single agent treatment (Cohorts A, B) or in combination with gemcitabine (Cohort C). All participants received the same dose in the respective Cohorts. The study was terminated due to the discontinuation of the overall development program of tusamitamab ravtansine by the Sponsor.
Groups:
- Cohort A: Metastatic Breast Cancer (mBC): Participants with mBC received an intravenous (IV) infusion of tusamitamab ravtansine at a loading dose of 170 milligram per square meter (mg/m^2) on Day 1 of Cycle 1 (cycle duration: 2 weeks), followed by 100 mg/m^2 every 2 weeks (Q2W) from Cycle 2 until documented disease progression, unacceptable toxicity, new anticancer therapy initiation, or the participant's or Investigator's decision to stop the treatment.
- Cohort B: Metastatic Pancreatic Adenocarcinoma (mPAC): Participants with mPAC received an IV infusion of tusamitamab ravtansine at a loading dose of 170 mg/m^2 on Day 1 of Cycle 1 (cycle duration: 2 weeks), followed by 100 mg/m^2 Q2W from Cycle 2 until documented disease progression, unacceptable toxicity, new anticancer therapy initiation, or the participant's or Investigator's decision to stop the treatment.
- Cohort C: Metastatic Pancreatic Adenocarcinoma (mPAC): Participants with mPAC received an IV infusion of tusamitamab ravtansine at an initial loading dose of 170 mg/m^2 on Day 1, followed by 100 mg/m^2 Q2W along with gemcitabine 1000 mg/m^2 on Days 1, 8, and 15 every 4 weeks (Q4W) until documented disease progression, unacceptable toxicity, new anticancer therapy initiation, or the participant's or Investigator's decision to stop the treatment.
Period: Overall Study
Arm/Group | Cohort A: Metastatic Breast Cancer (mBC) | Cohort B: Metastatic Pancreatic Adenocarcinoma (mPAC) | Cohort C: Metastatic Pancreatic Adenocarcinoma (mPAC)
Started | 6 | 28 | 16
Completed | 6 | 23 | 13
Not Completed | 0 | 5 | 3
Not completed — Study terminated by sponsor | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 5 | 0
Not completed — Not related to Coronavirus disease 2019 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All-treated population included all enrolled participants exposed to the study treatment, regardless of the amount of treatment administered.
Groups:
- Cohort A: mBC: Participants with mBC received an IV infusion of tusamitamab ravtansine at a loading dose of 170 mg/m^2 on Day 1 of Cycle 1 (cycle duration: 2 weeks), followed by 100 mg/m^2 Q2W from Cycle 2 until documented disease progression, unacceptable toxicity, new anticancer therapy initiation, or the participant's or Investigator's decision to stop the treatment.
- Cohort B: mPAC: Participants with mPAC received an IV infusion of tusamitamab ravtansine at a loading dose of 170 mg/m^2 on Day 1 of Cycle 1 (cycle duration: 2 weeks), followed by 100 mg/m^2 Q2W from Cycle 2 until documented disease progression, unacceptable toxicity, new anticancer therapy initiation, or the participant's or Investigator's decision to stop the treatment.
- Cohort C: mPAC: Participants with mPAC received an IV infusion of tusamitamab ravtansine at an initial loading dose of 170 mg/m^2 on Day 1, followed by 100 mg/m^2 Q2W along with gemcitabine 1000 mg/m^2 on Days 1, 8, and 15 Q4W until documented disease progression, unacceptable toxicity, new anticancer therapy initiation, or the participant's or Investigator's decision to stop the treatment.
- Total: Total of all reporting groups
Arm/Group | Cohort A: mBC | Cohort B: mPAC | Cohort C: mPAC | Total
Number analyzed (Participants) | 6 | 28 | 16 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (7.3) | 63.8 (11.8) | 65.0 (7.9) | 62.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 18 | 7 | 31
  Male | 0 | 10 | 9 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 19 | 15 | 38
  Asian | 1 | 2 | 1 | 4
  Unknown | 0 | 4 | 0 | 4
  Not reported | 1 | 3 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. CR was defined as disappearance of all target and non-target lesions, and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeter (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From date of first study treatment administration (Day 1) up to maximum exposure of treatment: 26.1 weeks (Cohort A), 51.6 weeks (Cohort B), 43.3 weeks (Cohort C)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: mBC | Cohort B: mPAC | Cohort C: mPAC
Number analyzed (Participants) | 6 | 28 | 16
percentage of participants | 0 [0.00 to 45.93] | 3.6 [0.09 to 18.35] | 31.3 [11.02 to 58.66]

2. Primary Outcome: Cohort C (Part 1): Number of Participants With Dose Limiting Toxicities (DLTs)
Description: The following adverse events (AEs) that occurred during the first cycle of treatment, unless due to disease progression or to a cause obviously unrelated to study treatment, were considered DLTs:
  1. Hematological abnormalities: grade 4 neutropenia for 7 or more consecutive days, grade 3 to 4 neutropenia complicated by fever or microbiologically or radiographically documented infection, grade greater than or equal to (≥) 3 thrombocytopenia associated with clinically significant bleeding requiring clinical intervention;
  2. Non-hematological abnormalities: grade 4 non-hematologic AE, grade ≥3 keratopathy.
  In addition, any other AE that the recruiting Investigators and Sponsor deemed to be dose limiting, regardless of its grade, was also considered as DLT.
Time Frame: Cycle 1 (28 days)
Population: DLT-evaluable population (Cohort C Part 1) included participants who received 1 cycle with at least 80% of the intended dose for both tusamitamab ravtansine at each of the first 2 infusions and gemcitabine at each of the 3 first infusions unless they discontinued the study treatment before the end of Cycle 1 due to a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort C: mPAC
Number analyzed (Participants) | 3
Participants | 0

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. A serious adverse event was defined as any AE that, at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission of any infectious agent via an authorized medicinal product. TEAEs were defined as AEs that developed, worsened, or became serious during the treatment-emergent period (defined as the period from the first study treatment administration to the last study treatment administration + 30 days).
Time Frame: From date of first study treatment administration (Day 1) up to 30 days after the last dose of study treatment, approximately 86.6 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: mBC | Cohort B: mPAC | Cohort C: mPAC
Number analyzed (Participants) | 6 | 28 | 16
Participants
  TEAEs | 6 | 28 | 16
  TESAEs | 0 | 16 | 9

4. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Hematology/Coagulation and Clinical Chemistry
Description: Blood samples were collected to determine the abnormalities in hematology/coagulation and clinical chemistry. Abnormality criteria was assessed as per the National Cancer Institute Common Terminology Criteria for Adverse Events v5.0. Hematological and coagulation parameters assessed were white blood cells, platelets, neutrophils, lymphocytes, and international normalized ratio. Clinical chemistry parameters assessed were albumin, sodium, potassium, calcium, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, and total bilirubin. Only those categories in which at least 1 participant had >2 grade worsening in laboratory abnormalities are reported.
Time Frame: as for outcome 3
Population: All-treated population included all enrolled participants exposed to the study treatment, regardless of the amount of treatment administered. Only those participants with data collected for the specified category are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: mBC | Cohort B: mPAC | Cohort C: mPAC
Number analyzed (Participants) | 6 | 27 | 15
Participants
  White blood cell decreased: number analyzed (Participants) | 4 | 26 | 14
  White blood cell decreased | 0 | 1 | 0
  Platelet count decreased: number analyzed (Participants) | 5 | 22 | 11
  Platelet count decreased | 0 | 0 | 1
  Neutrophil count decreased: number analyzed (Participants) | 6 | 26 | 15
  Neutrophil count decreased | 0 | 1 | 2
  Lymphocyte count decreased: number analyzed (Participants) | 4 | 18 | 13
  Lymphocyte count decreased | 0 | 0 | 2
  International normalized ratio increased: number analyzed (Participants) | 6 | 24 | 14
  International normalized ratio increased | 0 | 1 | 1
  Hypoalbuminemia: number analyzed (Participants) | 6 | 24 | 12
  Hypoalbuminemia | 0 | 1 | 0
  Hyponatremia: number analyzed (Participants) | 5 | 21 | 13
  Hyponatremia | 0 | 3 | 1
  Hyperkalemia | 0 | 1 | 0
  Hypocalemia: number analyzed (Participants) | 4 | 23 | 14
  Hypocalemia | 0 | 2 | 0
  Hypercalemia: number analyzed (Participants) | 6 | 26 | 12
  Hypercalemia | 0 | 0 | 2
  Alanine aminotransferase increased: number analyzed (Participants) | 6 | 26 | 15
  Alanine aminotransferase increased | 0 | 1 | 2
  Aspartate aminotransferase increased: number analyzed (Participants) | 6 | 26 | 15
  Aspartate aminotransferase increased | 0 | 1 | 0
  Alkaline phosphatase increased: number analyzed (Participants) | 6 | 26 | 15
  Alkaline phosphatase increased | 0 | 1 | 0
  Total bilirubin increased: number analyzed (Participants) | 6 | 26 | 15
  Total bilirubin increased | 1 | 2 | 1

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of first tusamitamab ravtansine administration to the date of the first documented disease progression according to RECIST v1.1 or death due to any cause, whichever came first. Disease progression was defined as unequivocal progression of existing non-target lesions; at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: mBC | Cohort B: mPAC | Cohort C: mPAC
Number analyzed (Participants) | 6 | 28 | 16
months | 3.71 [1.314 to NA] — NA indicates that the upper limit of 95% confidence interval (CI) was not estimable due to insufficient number of participants with events | 1.87 [1.643 to 2.267] | 4.73 [1.873 to NA] — NA indicates that the upper limit of 95% CI was not estimable due to insufficient number of participants with events

6. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who achieved confirmed CR, confirmed PR or stable disease (SD) as per RECIST v1.1. CR was defined as disappearance of all target and non-target lesions, and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD was defined as neither sufficient shrinkage from the baseline study to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference the smallest sum of diameters while on study.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: mBC | Cohort B: mPAC | Cohort C: mPAC
Number analyzed (Participants) | 6 | 28 | 16
percentage of participants | 66.7 [22.28 to 95.67] | 28.6 [13.22 to 48.67] | 75.0 [47.62 to 92.73]

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from first documented evidence of confirmed CR or confirmed PR until progressive disease determined per RECIST v1.1 or death from any cause, whichever occurred first. CR was defined as disappearance of all target and non-target lesions, and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Disease progression was defined as unequivocal progression of existing non-target lesions; at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 1
Population: All-treated population included all enrolled participants exposed to the study treatment, regardless of the amount of treatment administered. Only participants with response are analyzed. None of the participants in Cohort A had confirmed CR or PR; hence DOR could not be derived.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: mBC | Cohort B: mPAC | Cohort C: mPAC
Number analyzed (Participants) | 0 | 1 | 5
months |  | 4.11 [NA to NA] — NA indicates that the upper and lower limit of 95% CI were not estimable due to insufficient number of participants with events. | 7.26 [3.713 to NA] — NA indicates that the upper limit of 95% CI was not estimable due to insufficient number of participants with events.

8. Secondary Outcome: Number of Participants With Treatment-emergent Anti-therapeutic Antibodies (ATAs) Against Tusamitamab Ravtansine
Description: Blood samples were collected for assessing the presence of ATA against tusamitamab ravtansine in plasma. The number of participants with treatment-emergent ATA i.e., either seroconverted (treatment-induced ATAs) or boosted their pre-existing ATA response (treatment-boosted ATAs) during the study are reported.
Time Frame: From date of first study treatment administration (Day 1) up to 30 days after the last dose of study treatment administration [maximum exposure of treatment: 26.1 weeks (Cohort A), 51.6 weeks (Cohort B), 43.3 weeks (Cohort C)]
Population: ATA population included all treated participants with at least 1 post-baseline ATA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: mBC | Cohort B: mPAC | Cohort C: mPAC
Number analyzed (Participants) | 6 | 21 | 4
Participants | 2 | 5 | 2

9. Secondary Outcome: Cohort C: Maximum Concentration Observed After Infusion (Cmax) of Tusamitamab Ravtansine
Description: Blood samples were collected for the measurement of Cmax of tusamitamab ravtansine. Cmax was calculated using non-compartmental method.
Time Frame: Cycle 1: Day 1: Start of infusion, end of infusion, 3, 72, 168, and 336 hours post-start of infusion (cycle duration: 28 days)
Population: Pharmacokinetic (PK) population included all treated participants with at least 1 post-baseline PK result with adequate documentation of dosing and sampling dates and times.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Cohort C: mPAC
Number analyzed (Participants) | 8
microgram per milliliter (mcg/mL) | 88.3 (17.8)

10. Secondary Outcome: Cohort C: Area Under the Plasma Concentration Versus Time Curve Calculated Using the Trapezoidal Method From Time 0 to 14 Days (AUC0-14d) of Tusamitamab Ravtansine
Description: Blood samples were collected for the measurement of AUC0-14d of tusamitamab ravtansine. AUC0-14d was calculated using non-compartmental method.
Time Frame: as for outcome 9
Population: PK population included all treated participants with at least 1 post-baseline PK result with adequate documentation of dosing and sampling dates and times. Only those participants with data collected for this outcome measure are reported.
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Cohort C: mPAC
Number analyzed (Participants) | 7
day*mcg/mL | 473 (85.7)

11. Secondary Outcome: Cohort C: Total Body Clearance From Plasma (CL) of Gemcitabine
Description: Blood samples were collected for the measurement of CL of gemcitabine. CL was calculated using non-compartmental method.
Time Frame: Cycle 1: Days 1 and 8: Start of infusion, end of infusion, 0.25, 1, 1.5, and 2 hours post-start of infusion (cycle duration: 28 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Cohort C: mPAC
Number analyzed (Participants) | 3
liter per hour | 169 (93.8)

12. Secondary Outcome: Cohort C: Cmax of Gemcitabine Metabolite (dFdU)
Description: Blood samples were collected for the measurement of Cmax of dFdU. Cmax was calculated using non-compartmental method.
Time Frame: as for outcome 11
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort C: mPAC
Number analyzed (Participants) | 3
mcg/mL | 31.4 (7.27)

ADVERSE EVENTS:
Time Frame: From date of first study treatment administration (Day 1) up to 30 days after the last dose of study treatment, approximately 86.6 weeks.
Description: Analysis was performed on all-treated population.
Arm/Group | Cohort A: mBC | Cohort B: mPAC | Cohort C: mPAC
All-Cause Mortality (participants affected / at risk) | 4/6 | 21/28 | 9/16
Serious Adverse Events (participants affected / at risk) | 0/6 | 16/28 | 9/16
Other Adverse Events (participants affected / at risk) | 6/6 | 23/28 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: mBC (N=6) | Cohort B: mPAC (N=28) | Cohort C: mPAC (N=16)
Biliary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea Infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Aspiration (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal Stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric Dilatation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis Erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary Obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice Cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Complication Associated With Device (General disorders) | 0 (0) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 0 (0) | 6 (6) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Radiation Osteitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: mBC (N=6) | Cohort B: mPAC (N=28) | Cohort C: mPAC (N=16)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Candida Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (5)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 4 (5)
Contrast Media Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Contrast Media Reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 9 (10) | 5 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Iron Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Diabetic Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 1 (2) | 4 (5)
Eye Pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (2) | 2 (2) | 0 (0)
Keratopathy (Eye disorders) | 1 (1) | 5 (5) | 2 (3)
Vision Blurred (Eye disorders) | 1 (1) | 1 (1) | 3 (3)
Xerophthalmia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 7 (8) | 3 (4)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 5 (7) | 3 (5)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Gastrointestinal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (6) | 4 (4) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (5) | 2 (5) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 4 (4)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 13 (15) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2) | 4 (4)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 2 (4)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 4 (4) | 2 (2)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram Qt Prolonged (Investigations) | 0 (0) | 2 (2) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 2 (6)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (4)
Platelet Count Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 4 (4) | 1 (3)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated due to the discontinuation of the overall development program of tusamitamab ravtansine (SAR408701) by the Sponsor on 20 December 2023.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT04659603/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT04659603/SAP_001.pdf